CLINICAL TRIAL: NCT04962698
Title: Robotically Augmented Mental Practice for Neuromotor Facilitation
Brief Title: Robotically Augmented Mental Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H21154; R21NS118435 (NIH)
Record Dates: First submitted 2021-07-02; First posted 2021-07-15 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Hand; Imagery; Robot
MeSH Terms: conditions — Stroke | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Participants in a single group will receive various types of interventions in random order. The types of interventions are the same across subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy participants (Experimental): All participants will receive seven types of interventions in random order. The types of interventions are the same across subjects.
  Interventions: Behavioral: Visual motor imagery (MI); Behavioral: Kinesthetic MI; Behavioral: Robotic-Hand Interaction with MI; Behavioral: Robotic-Hand Interaction without MI; Behavioral: Virtual-Hand Interaction; Behavioral: Robotic Action Observation; Behavioral: Rest
- Post-Stroke participants (Experimental): All participants will receive three types of interventions in random order. The types of interventions are the same across subjects.
  Interventions: Behavioral: Visual motor imagery (MI); Behavioral: Robotic-Hand Interaction with MI; Behavioral: Rest

INTERVENTIONS:
Behavioral: Visual motor imagery (MI) — Subjects will relax their muscles and perform conventional visual motor imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
Behavioral: Kinesthetic MI — The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Arms: Healthy participants
Behavioral: Robotic-Hand Interaction with MI — Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
Behavioral: Robotic-Hand Interaction without MI — Subjects will perform the Robot-Hand Interaction without MI.
  Arms: Healthy participants
Behavioral: Virtual-Hand Interaction — Subjects will interact with visual feedback of virtual robot actions on a monitor.
  Arms: Healthy participants
Behavioral: Robotic Action Observation — Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Arms: Healthy participants
Behavioral: Rest — Subjects will rest without a task.

SUMMARY:
This project will develop and test a new paradigm of motor imagery for facilitating neuromotor excitability and performance of distal muscles in the upper limb by adopting a robotic prosthesis and integrating proven procedures for neuromotor facilitation. The scientific purpose of the study is to understand the effect of controlling a detached robotic prosthesis with proximal muscle activation on brain excitability of the resting arm muscles as well as reaction time. The efficacy of this task will be understood by comparing with other task conditions (motor imagery only, 2D visual feedback on a monitor, etc.) that do not involve the robotic prosthesis. The test of the developed system will be performed in healthy able-bodied adults. The feasibility of the system will be examined in post-stroke adults.

DETAILED DESCRIPTION:
This study consists of experiments on two non-consecutive days in the Human Neuromuscular Physiology Laboratory located in the Biological Sciences/Applied Physiology Building of Georgia Tech. If subjects qualify and agree to take part in this study, subjects will be asked to read and sign the consent form. The whole procedure will last about 3 hours per day, including preparation. Subjects will come to the lab on two separate days on the same tasks. The first day will serve as familiarization with the same tasks as the second day. Subjects will perform the following experiment. Individuals will sit upright and relax their hands and shoulders. The right hand and forearm will be rested on a plate hidden below a table. The robotic hand will be placed on the table as one would normally place own arm on the table. There will be no physical connection between the hand and the robotic hand. Subjects will activate the abdominal muscles for making a grasping movement of the robotic hand. For making a releasing movement of the robotic hand, subjects will activate the back muscles. Muscle activity will be recorded with two small sensors on each muscle. Subjects will practice activation of each muscle while watching the signal on a monitor. In each muscle, a clearer signal will be used for controlling the robotic digits. Healthy subjects only: Healthy subjects will perform the following tasks A-F. [A: Rest] Subjects will relax the muscles without physical or cognitive effort while gazing at the turned-off monitor. [B: Robotic action observation] Subjects will relax the muscles and focus on observing the computer-controlled grasp and release actions (2 s in each movement) of the robotic prosthesis. [C: Visual MI] Subjects will relax the muscles and perform conventional visual motor imagery (MI). With the guidance of audio instruction, the subjects will image the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction. [D: Kinesthetic MI] The same MI procedure as Task C will be performed, except that the subjects will focus on the kinesthetic sensation that was felt with the imaged motions. [E: Robotic-Hand Interaction with MI] Subjects will perform robotically augmented mental practice (see below detailed description) for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also image the kinesthetic sensation that was felt with the corresponding motions with the right arm. [F: Virtual-Hand Interaction robot] Subjects will perform Task E with visual feedback of virtual robot actions in 2D on a monitor. [G: Robotic-Hand Interaction without MI] Subjects will perform Task E without MI. As a reaction task, subjects will flex the index finger as soon as they hear an auditory cue. Post-stroke subjects only: Tasks C [Visual MI], E [Robotic-Hand Interaction with MI], and A [Rest] above will be performed by post-stroke subjects with right-side hemiparesis who can volitionally activate fingers and proximal muscles. As a reaction task, subjects will flex the index finger as soon as an auditory cue is heard. TMS (both healthy and post-stroke subjects): During the above-mentioned tasks, brain stimulation (called TMS) will be applied over the motor cortex in the left hemisphere. The TMS procedure will follow the one used in the previous studies by the investigators. A TMS coil will be placed over a precise point on the scalp where the investigators will stimulate the brain to make the muscle move. The investigators will tell the subject when the stimulation portion of the procedure is about to begin. The first part of the procedure will be to find the area of the brain that controls muscles. These investigators will position the TMS coil on the head and will give the subject a series of stimulations (called magnetic pulses). Once the spot that controls the muscles is identified, the investigators will find the least amount of stimulation needed to activate the resting muscles. The second part of the procedure will be to evoke muscle contraction with TMS at rest and during the tasks described above. The investigators will apply TMS with 5-second intervals or more. Robotically augmented practice (Task E and F above): An individual will use proximal muscle contractions to flex and extend the robotic prosthesis digits for performing a grasp-release task. 1) Grasp. The individual will activate the proximal muscles as if for a retrieving motion (the back muscles) for 2 s. This muscle activation controls the robotic hand to flex the digits to grasp a cylinder-shaped object. 2) Release. The individual will relax the above-activated proximal muscles and activate the proximal muscles as if for a reaching motion (the abdominal muscles) for 2 s. This muscle activation controls the robotic hand to extend the digits to release the object. After releasing the object, the individual will relax the proximal muscles. The individual will repeat this sequence while observing and hearing the actions of the robotic hand.

ELIGIBILITY:
Inclusion Criteria for Healthy able-bodied volunteers:

* 18-39 years old, men and women

Inclusion Criteria for Right-handed Post-stroke adults:

* 21-75 years old
* Right-handed
* Longer than 6 months post-stroke
* Persistent hemiparesis on the right upper extremity (UE)
* Residual UE voluntary movement as indicated by a score of 1-3 on the motor arm item of the NIH Stroke Scale (NIHSS) and a score of 19-55 on the UE portions of the Fugl Meyer Assessment (UE-FMA)
* Preserved cognitive function
* Ability to follow and read simple instructions as indicated by a score of 1 or above on item #9 on the best language items of the NIHSS

Exclusion Criteria for both healthy and post-stroke individuals: To ensure the safety associated with TMS, the following adults will be excluded (*, not applicable to post-stroke subjects):

* Had an adverse reaction to TMS. Had epilepsy or seizure.
* Have any implanted devices such as a neurostimulator or cochlear implant.
* Had a stroke or lesion (including tumor) in your brain*. Had a head injury or brain surgery*.
* Suffer from frequent or severe headaches.
* Had a fainting spell or syncope.
* Have any metal in the head such as shrapnel, surgical clips, or fragments from welding or metalwork.
* Have any implanted device such as cardiac pacemakers, medical pumps, or intra-cardiac lines.
* Had any brain-related conditions*.
* Had any illness that caused brain injury* (i.e. meningitis, aneurysm, brain tumor).
* Had any head trauma that was associated with a loss of consciousness or diagnosed as a concussion.
* Being treated for any psychiatric condition (i.e. depression, anxiety, PTSD, schizophrenia).
* Had more than 2 cups of coffee/caffeinated beverages in the last 12 hours.
* Had more than 2 alcoholic beverages in the last 12 hours.
* Had less than 6 hours of sleep in the last 24 hours.
* Suspected of pregnancy.

Additional Exclusion Criteria for post-stroke adults:

* A first stroke less than 6 months or more than 24 months prior to the participation.
* Hemiparesis on the left side.
* Hemorrhagic stroke.
* Cerebellar stroke.
* Severe sensory impairment as indicated by the score of 2 (Severe to total sensory loss; the patient is not aware of being touched in the face, arm, and leg) in item #8 (Sensory) of the NIH Stroke Scale (NIHSS).
* Serious uncontrolled medical conditions.
* Severe apraxia of speech.
* Excessive pain in any joint of the more affected extremity that could limit the ability to cooperate with the intervention, as judged by the examining clinician.
* Receiving any anti-spasticity drugs orally at the time of expected participation, 3 months prior, or wish to or is scheduled to receive injections prior to study completion.
* Received phenol injections less than 12 months prior to receiving therapy.
* Unable to stand independently for 2 min., transfer independently to and from the toilet, or perform sit-to-stand.
* A score of less than 24 on the Folstein Mini-Mental State Examination.
* Passive range of motion less than 45 degrees for abduction, flexion or external rotation at the shoulder, or pronation of forearm; or greater than 30 degrees flexion contracture at any finger joint.
* Active range of motion less than 10 degrees for finger flexion or extension.
* Inability to volitionally activate right UE proximal muscles used for EMG placement.
* Clinical judgment of a) a major medical disorder that substantially reduces the likelihood that a subject will be able to comply with all study procedures, b) unable to successfully perform all rehabilitation exercise test examples, or c) unable or unwilling to perform study procedures/therapy, or expectation of non-compliance with study procedures/therapy.
* No TMS response in the first dorsal interosseous muscle in the right hand.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minoru Shinohara, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Human Neuromuscular Physiology Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: (Cross-over design but presented as a single group because of many sequences)
  All participants will receive seven types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery: Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Kinesthetic MI: The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Robotic-hand interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Robotic-hand interaction without MI: Subjects will perform the robotically augmented practice without MI.
  Virtual-hand interaction: Subjects will perform the augmented practice with visual feedback of virtual robot actions on a monitor.
  Robotic action observation: Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Rest: Subjects will rest without a task.
- Post-Stroke Participants: All participants will receive three types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery: Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Robotic-hand interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Rest: Subjects will rest without a task.
Period: Motor Imagery
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 6
Completed | 18 | 4
Not Completed | 1 | 2
Not completed — Technical difficulty | 1 | 0
Not completed — Exclusion criteria met after enrollment | 0 | 2
Period: Kinesthetic MI
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 0
Completed | 18 | 0
Not Completed | 1 | 0
Not completed — Technical difficulty | 1 | 0
Period: Robotic-hand Interaction With MI
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 6
Completed | 18 | 4
Not Completed | 1 | 2
Not completed — Technical difficulty | 1 | 0
Not completed — Exclusion criteria met after enrollment | 0 | 2
Period: Robotic-hand Interaction Without MI
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 0
Completed | 18 | 0
Not Completed | 1 | 0
Not completed — Technical difficulty | 1 | 0
Period: Virtual-hand Interaction
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 0
Completed | 18 | 0
Not Completed | 1 | 0
Not completed — Technical difficulty | 1 | 0
Period: Robotic Action Observation
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 0
Completed | 18 | 0
Not Completed | 1 | 0
Not completed — Technical difficulty | 1 | 0
Period: Rest
Arm/Group | Healthy Participants | Post-Stroke Participants
Started | 19 | 6
Completed | 18 | 4
Not Completed | 1 | 2
Not completed — Technical difficulty | 1 | 0
Not completed — Exclusion criteria met after enrollment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Healthy Participants: All participants will receive various types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery (MI): Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Kinesthetic MI: The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Robotic-hand interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Robotic-hand interaction without MI: Subjects will perform the robotically augmented practice without MI.
  Virtual-hand interaction: Subjects will perform the augmented practice with visual feedback of virtual robot actions on a monitor.
  Robotic action observation: Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Rest: Subjects will rest without a task.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Post-Stroke Participants | Total
Number analyzed (Participants) | 19 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 6 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 17 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 7 | 5 | 12
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: MEP Amplitude
Description: Peak-to-peak amplitude of motor evoked potential (MEP) of the hand muscle
Time Frame: 1 day
Population: Post-stroke data were not included in the overall statistical tests because they have distinct neuromotor characteristics and cannot be mixed with healthy samples. Post-stroke data were not statistically tested independently either because the number of subjects is too small to achieve appropriate statistical power. This strategy was as originally planned.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Healthy Participants: All participants will receive seven types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery (MI): Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Kinesthetic MI: The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Robotic-Hand Interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Robotic-Hand Interaction without MI: Subjects will perform the Robot-Hand Interaction without MI.
  Virtual-Hand Interaction: Subjects will interact with visual feedback of virtual robot actions on a monitor.
  Robotic action observation: Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Rest: Subjects will rest without a task.
- Post-Stroke Participants: All participants will receive three types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery (MI): Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Robotic-Hand Interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Rest: Subjects will rest without a task.
Arm/Group | Healthy Participants | Post-Stroke Participants
Number analyzed (Participants) | 18 | 4
mV
  Motor Imagery | 0.813 (0.800) | 0.475 (0.300)
  Kinesthetic Motor Imagery: number analyzed (Participants) | 18 | 0
  Kinesthetic Motor Imagery | 0.916 (0.695) |
  Robotic-Hand Interaction with MI | 1.237 (1.010) | 0.451 (0.307)
  Robotic-Hand Interaction without MI: number analyzed (Participants) | 18 | 0
  Robotic-Hand Interaction without MI | 1.019 (0.823) |
  Virtual-Hand Interaction: number analyzed (Participants) | 18 | 0
  Virtual-Hand Interaction | 1.197 (1.010) |
  Robotic Action Observation: number analyzed (Participants) | 18 | 0
  Robotic Action Observation | 0.899 (0.652) |
  Rest | 1.106 (0.715) | 0.810 (0.567)
Statistical Analysis 1: Comparison: Healthy Participants; Test type: Superiority; p > 0.00238, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was 0.00238, which was adjusted from the original 0.05 as described below; The alpha value for p-value comparison was adjusted for 21 pair-wise comparisons (0.05/21 = 0.00238) across seven tasks

2. Primary Outcome: Reaction Time
Description: Reaction time of the index finger in response to an auditory cue (reaction time test)
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Helathy Participants: All participants will receive seven types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery (MI): Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Kinesthetic MI: The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Robotic-Hand Interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Robotic-Hand Interaction without MI: Subjects will perform the Robot-Hand Interaction without MI.
  Virtual-Hand Interaction: Subjects will interact with visual feedback of virtual robot actions on a monitor.
  Robotic action observation: Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Rest: Subjects will rest without a task.
Arm/Group | Helathy Participants | Post-Stroke Participants
Number analyzed (Participants) | 18 | 4
ms
  Motor Imagery | 293.6 (43.0) | 522.0 (205.4)
  Kinesthetic Motor Imagery: number analyzed (Participants) | 18 | 0
  Kinesthetic Motor Imagery | 286.4 (57.5) |
  Robotic-Hand Interaction with MI | 275.7 (51.5) | 378.6 (107.0)
  Robotic-Hand Interaction without MI: number analyzed (Participants) | 18 | 0
  Robotic-Hand Interaction without MI | 271.7 (38.3) |
  Virtual-Hand Interaction: number analyzed (Participants) | 18 | 0
  Virtual-Hand Interaction | 273.4 (44.2) |
  Robotic Action Observation: number analyzed (Participants) | 18 | 0
  Robotic Action Observation | 259.9 (38.2) |
  Rest | 234.2 (38.7) | 362.8 (94.4)
Statistical Analysis 1: Comparison: Helathy Participants; Test type: Superiority; p < 0.001, ANOVA — The threshold for statistical significance was 0.05

3. Primary Outcome: Peak EMG
Description: Peak EMG amplitude of the hand muscle during the reaction time test was determined in each intervention. After identifying the maximal peak EMG value among the interventions, peak EMG value in each task was normalized to that maximal peak EMG, expressed as the ratio.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Healthy Participants | Post-Stroke Participants
Number analyzed (Participants) | 18 | 4
Ratio
  Motor Imagery | 0.602 (0.292) | 0.517 (0.320)
  Kinesthetic Motor Imagery: number analyzed (Participants) | 18 | 0
  Kinesthetic Motor Imagery | 0.602 (0.277) |
  Robotic-Hand Interaction with MI | 0.721 (0.290) | 0.954 (0.093)
  Robotic-Hand Interaction without MI: number analyzed (Participants) | 18 | 0
  Robotic-Hand Interaction without MI | 0.699 (0.311) |
  Virtual-Hand Interaction: number analyzed (Participants) | 18 | 0
  Virtual-Hand Interaction | 0.683 (0.302) |
  Robotic Action Observation: number analyzed (Participants) | 18 | 0
  Robotic Action Observation | 0.488 (0.288) |
  Rest | 0.530 (0.256) | 0.599 (0.313)
Statistical Analysis 1: Comparison: Healthy Participants; Test type: Superiority; p = 0.028, ANOVA — The threshold for statistical significance was 0.05

4. Primary Outcome: Maximal Rate of Force Development
Description: Maximal rate of force development during a reaction time test
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: N/s
Arm/Group | Healthy Participants | Post-Stroke Participants
Number analyzed (Participants) | 18 | 4
N/s
  Motor Imagery | 44.0 (39.8) | 12.6 (6.7)
  Kinesthetic Motor Imagery: number analyzed (Participants) | 18 | 0
  Kinesthetic Motor Imagery | 42.9 (33.0) |
  Robotic-Hand Interaction with MI | 56.7 (53.9) | 23.0 (15.9)
  Robotic-Hand Interaction without MI: number analyzed (Participants) | 18 | 0
  Robotic-Hand Interaction without MI | 61.6 (61.5) |
  Virtual-Hand Interaction: number analyzed (Participants) | 18 | 0
  Virtual-Hand Interaction | 57.0 (57.3) |
  Robotic Action Observation: number analyzed (Participants) | 18 | 0
  Robotic Action Observation | 39.1 (33.2) |
  Rest | 40.8 (48.1) | 20.0 (15.4)
Statistical Analysis 1: Comparison: Healthy Participants; Test type: Superiority; p < 0.00231, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was 0.00238, which was adjusted from the original 0.05 as described below; The alpha value for p-value comparison was adjusted for 21 pair-wise comparisons (0.05/21 = 0.00238) across seven tasks

5. Primary Outcome: Peak Force
Description: Peak force of the index finger during a reaction time test
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: N
Arm/Group | Healthy Participants | Post-Stroke Participants
Number analyzed (Participants) | 18 | 4
N
  Motor Imagery | 4.369 (4.018) | 1.968 (1.869)
  Kinesthetic Motor Imagery: number analyzed (Participants) | 18 | 0
  Kinesthetic Motor Imagery | 4.370 (4.010) |
  Robotic-Hand Interaction with MI | 5.342 (5.557) | 3.708 (3.378)
  Robotic-Hand Interaction without MI: number analyzed (Participants) | 18 | 0
  Robotic-Hand Interaction without MI | 5.666 (5.553) |
  Virtual-Hand Interaction: number analyzed (Participants) | 18 | 0
  Virtual-Hand Interaction | 5.105 (5.464) |
  Robotic Action Observation: number analyzed (Participants) | 18 | 0
  Robotic Action Observation | 3.741 (3.385) |
  Rest | 3.537 (3.878) | 3.312 (4.107)
Statistical Analysis 1: Comparison: Healthy Participants; Test type: Superiority; p < 0.0020, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was 0.00238, which was adjusted from the original 0.05 as described below; The alpha value for p-value comparison was adjusted for 21 pair-wise comparisons (0.05/21 = 0.00238) across seven tasks

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Healthy Participants: All participants will receive various types of interventions in random order. The types of interventions are the same across subjects.
  Visual motor imagery (MI): Subjects will relax their muscles and perform conventional visual mental imagery (MI). With the guidance of audio instruction, the subjects will imagine the grasp and release motions with the right arm for 2 s in each motion in their mind. There will be no proximal muscle contraction.
  Kinesthetic MI: The same MI procedure as Visual MI will be performed, except that the subjects will focus on the kinesthetic sensation that they would feel with the imagined motions.
  Robotic-hand interaction with MI: Subjects will perform robotically augmented mental practice for grasp and release motions with the activation control of the proximal muscles. During this task, subjects will also imagine the kinesthetic sensation that they would feel with the corresponding motions with the right arm.
  Robotic-hand interaction: Subjects will perform the robotically augmented practice without MI.
  Virtual-hand interaction: Subjects will perform the augmented practice with visual feedback of virtual robot actions on a monitor.
  Robotic action observation: Subjects will relax their muscles and focus on observing the computer-controlled grasp and release actions of the robotic hand.
  Rest: Subjects will rest without a task.
Arm/Group | Healthy Participants | Post-Stroke Participants
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/6
Other Adverse Events (participants affected / at risk) | 0/19 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT04962698/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04962698/ICF_002.pdf